CLINICAL TRIAL: NCT03972319
Title: Omega-3 Supplementation for LIver VolumE Reduction Study (OLIVER) Study
Acronym: OLIVER
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khoo Teck Puat Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OLIVER 1.3
Record Dates: First submitted 2019-05-28; First posted 2019-06-03 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Fatty Liver; Bariatric Surgery Candidate
Keywords: omega 3; bariatric surgery; fatty liver; vlcd
MeSH Terms: conditions — Fatty Liver | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omega-3 Supplementation (Experimental): Proof of Concept and Safety Study of 4 weeks of Omega-3 supplementation pre- Bariatric Surgery
  Interventions: Dietary Supplement: 2 capsules of Concentrated omega-3 triglycerides- fish 1000mg (600mg Eicosapentaenoic acid (EPA), 1400mg Docosahexaenoic acid (DHA)) per day

INTERVENTIONS:
Dietary Supplement: 2 capsules of Concentrated omega-3 triglycerides- fish 1000mg (600mg Eicosapentaenoic acid (EPA), 1400mg Docosahexaenoic acid (DHA)) per day — 4 weeks course of Omega-3 (2 capsules of Blackmores Omega Daily Concentrated Fish Oil per day

SUMMARY:
Omega-3 has been postulated to reduce hepatic steatosis by reducing lipogenic gene expression, exerting anti- inflammation action, reducing oxidative stress and improving glycemic control.

A recent meta-analysis by Parker et al.[1] found that omega-3 supplementation is associated with improvement in liver fat content as well as on Aspartate Aminotransferase (AST) levels. Omega-3 supplementation has also found to be useful in reducing blood triglyceride levels [2].

Recent studies by Iannelli et al. (2013) and Abidin et al.(2017) have also found that a 1 month supplementation of 1.5g/day and 2g/day of omega-3 supplementation resulted in reduced hepatic volume of 20% and 34.88 cm3 respectively.

The investigator's hypothesis is that a 4 weeks course of Omega-3 (2 capsules of Blackmores Omega Daily Concentrated Fish Oil per day; Each capsule Concentrated omega-3 triglycerides- fish 1000mg containing Omega-3 Marine Triglycerides 600mg as: 360mg Eicosapentaenoic acid (EPA), 240mg Docosahexaenoic acid (DHA)) taken as supplement, without any other dietary intervention pre Bariatric Surgery decreases significantly liver volume and facilitate access during surgery. And that shrinkage of liver volume also translates to improve biochemical parameters of fatty liver disease

DETAILED DESCRIPTION:
A total of 50 subjects booked for Bariatric Surgery with BMI up 45 will be recruited. Patients with pre-existing liver disease, excessive alcohol consumption and significant central obesity will be excluded.

Ultrasound examination of the liver with liver volume measurement, and blood tests, including Liver Function Tests (LFT) and platelet counts,is performed as part of the pre surgery work up.

The subjects are then given 4 weeks of Omega-3 supplements (2 capsules of Blackmores Omega Daily Concentrated Fish Oil per day: Concentrated omega-3 triglycerides- fish 1000mg (600mg Eicosapentaenoic acid (EPA), 1400mg Docosahexaenoic acid (DHA)).

Just before Surgery, a repeat of ultrasound examination and measurement of liver volume is carried out, as well as a repeat liver panel and platelet count.The subjects will have their weight and body composition recorded as well at this time.

At the time of the surgery, the surgeon makes a subjective assessment of the left lobe liver volume on a scale of 1 to 5, 5 being the largest. Additionally,ease of access to area under the left lobe of the liver is also subjectively assessed, on a scale of 1 to5, 5 being the most difficult.

ELIGIBILITY:
Inclusion Criteria:

* Subjects qualifying and scheduled for Bariatric Surgery (as according to Singapore Health Promotion Board- Ministry of Health Obesity Clinical Practice GuidelineJune 2016)
* BMI <45 with no significant central obesity.
* Has no pre-existing liver disease, or excess alcohol consumption.

Exclusion Criteria:

* Pre-existing liver disease
* Excessive alcohol consumption
* Prior history of allergy to omega-3 products, salmon or other- related products
* central obesity
* Pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Changes of Liver Volume Facilitating Access during Bariatric Surgery | After 4 weeks of Omega-3 supplement
  To demonstrate that Omega-3 oil taken as supplement, without any other dietary intervention pre Bariatric Surgery significantly changes liver volume and facilitates access during surgery.

SECONDARY OUTCOMES:
Change in Biochemical parameters (serum ALT levels) of fatty liver disease | After 4 weeks of Omega-3 supplement
  To demonstrate changes in liver volume also translates to improved biochemical parameters (serum Alanine Aminotransferase levels) of fatty liver disease.
Change in Biochemical parameters (serum AST levels) of fatty liver disease | After 4 weeks of Omega-3 supplement
  To demonstrate changes in liver volume also translates to improved biochemical parameters (serum Aspartate Aminotransferase levels) of fatty liver disease.
Change in Biochemical parameters (serum Platelet levels) of fatty liver disease | After 4 weeks of Omega-3 supplement
  To demonstrate changes in liver volume also translates to improved biochemical parameters (serum Platelet levels) of fatty liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Cheng, MBBS FRCS, Principal Investigator — Khoo Teck Puat Hospital; Deborah Ng, MBBS MMed, Principal Investigator — Khoo Teck Puat Hospital; Tan Chun Hai, MBBS FRCS, Study Director — Khoo Teck Puat Hospital; Lim Kheng Tian, MBBS FRCS, Study Director — Khoo Teck Puat Hospital; Tan Bo Chuan, MBBS FRCS, Study Director — Khoo Teck Puat Hospital; Babu Suresh Balasubramaniam, MBBS FRCR, Study Director — Khoo Teck Puat Hospital
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iannelli A, Martini F, Schneck AS, Ghavami B, Baudin G, Anty R, Gugenheim J. Preoperative 4-week supplementation with omega-3 polyunsaturated fatty acids reduces liver volume and facilitates bariatric surgery in morbidly obese patients. Obes Surg. 2013 Nov;23(11):1761-5. doi: 10.1007/s11695-013-0942-y. PMID 23686653
- See also: A randomised controlled trial comparing the use of omega-3 polyunsaturated fatty acid supplements versus very low calorie dietary restriction in obese Malaysian patients awaiting bariatric surgery — http://ales.amegroups.com/article/download/4052/4885